CLINICAL TRIAL: NCT07176832
Title: Bioavailability Study of Stiripentol After Single Oral Administration of Two Different Formulations (Capsule and Oral Suspension) in 24 Healthy Subjects
Brief Title: Bioavailability of Stiripentol After Single Oral Dose of Capsule vs Suspension in Healthy Subjects (STILIQ)
Acronym: STILIQ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocodex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STILIQ - STP 218; 2024-520103-38-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-29; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Dravet Syndrome; Epilepsy; Childhood; Epileptic Encephalopathy; Pediatric Epilepsy
Keywords: Stiripentol; Diacomit; Oral Suspension; Bioavailability; Pharmacokinetics; Antiepileptic Drug; Crossover Study; Healthy Volunteers; Pediatric Epilepsy; Dravet Syndrome Treatment
MeSH Terms: conditions — Epilepsies, Myoclonic; Epilepsy | interventions — stiripentol; Suspensions

STUDY DESIGN:
Intervention Model Description: A single center, two-way, 2 periods, open-label, cross-over, and randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A : Stiripentol Capsule then Oral Suspension (Experimental): Subjects randomized to Sequence A will receive a single oral dose of 1,000 mg stiripentol (2 × 500 mg capsules, Diacomit®) at the end of breakfast under fed conditions in Period 1, followed by a single oral dose of 1,000 mg stiripentol (20 mL oral suspension, 50 mg/mL, Diacomit®) in Period 2 after a 7-15 day
  Interventions: Drug: Stiripentol capsule (Diacomit®); Drug: Stiripentol oral suspension (Diacomit®)
- Sequence B : Stiripentol Oral Suspension then Capsule (Experimental): Subjects randomized to Sequence B will receive a single oral dose of 1,000 mg stiripentol (20 mL oral suspension, 50 mg/mL, Diacomit®) at the end of breakfast under fed conditions in Period 1, followed by a single oral dose of 1,000 mg stiripentol (2 × 500 mg capsules, Diacomit®) in Period 2 after a 7-15 day washout.
  Interventions: Drug: Stiripentol capsule (Diacomit®); Drug: Stiripentol oral suspension (Diacomit®)

INTERVENTIONS:
Drug: Stiripentol capsule (Diacomit®) — Single oral administration of 1,000 mg stiripentol (2 × 500 mg capsules) at the end of breakfast.
  Other Names: Stiripentol 500 mg capsule; Diacomit® capsule
Drug: Stiripentol oral suspension (Diacomit®) — Single oral administration of 1,000 mg stiripentol (20 mL oral suspension, 50 mg/mL) at the end of breakfast.
  Other Names: Stiripentol 50 mg/mL suspension; Diacomit® oral suspension

SUMMARY:
This is a Phase I, open-label, randomized, single-center, two-way cross-over study evaluating the relative bioavailability, pharmacokinetics, safety, and palatability of two formulations of stiripentol (Diacomit®), indicated in Dravet syndrome. The investigational products are 500 mg capsules (reference) and a 50 mg/mL oral suspension (test).

The primary objective is to compare the relative bioavailability of the two formulations after a single 1,000 mg oral dose under fed conditions, based on Cmax, AUC0-t, and AUC0-∞. Secondary objectives include other PK parameters (tmax, tlag, ke, t1/2) and characterization of metabolites MIa and MIb. Palatability of the suspension will be assessed by questionnaire.

Safety evaluation will include adverse events, laboratory tests, ECGs, urinalysis, drug and alcohol screening, serology, and vital signs.

Twenty-four healthy volunteers (18-50 years) will be enrolled. Eligibility: BMI 18-30 kg/m², weight ≥50 kg, normal ECG and labs, and informed consent. Women of childbearing potential must use effective contraception and test negative for pregnancy. Exclusions: significant disease, recent surgery or blood donation, hypersensitivity, difficulty swallowing, use of CYP modulators (e.g., carbamazepine, grapefruit, herbal products), drug or alcohol abuse, smoking >5 cigarettes/day, or inability to follow dietary restrictions. Subjects testing positive for HIV, HBV, HCV, or drugs of abuse will also be excluded.

Each participant will attend a screening visit within 28 days before dosing, then two 3-day hospitalizations separated by a 7-15-day washout. On Day 1 of each period, they will receive either two capsules (1,000 mg) or 20 mL suspension (1,000 mg). Blood will be collected at 36 timepoints (≈180 mL total) for PK assessment.

The total study duration per subject is about seven weeks, including screening, hospitalization, dosing, washout, and follow-up. Treatment consists of one dosing day per period.

Sample size was based on prior data: 21 pairs provide 80% power for bioequivalence within 0.80-1.25 bounds; 24 subjects will be recruited to account for dropouts. Analyses will include the Safety Set, PK Concentrations Set, and PK Analysis Set.

This trial aims to establish whether the oral suspension provides a PK profile comparable to capsules, while generating safety, tolerability, and palatability data to support a more convenient formulation for Dravet syndrome patients.

DETAILED DESCRIPTION:
Stiripentol (Diacomit®) is currently marketed in two dosage forms: capsules (250 and 500 mg) and powder for oral suspension in sachets (250 and 500 mg). The powder formulation was developed for patients unable to swallow capsules. A previous study in healthy volunteers demonstrated that the capsule and sachet formulations were bioequivalent in terms of AUC but not Cmax. The Cmax of the sachet formulation was approximately 23% higher than that of the capsule, outside the accepted bioequivalence range. As a result, clinical supervision is recommended when switching between capsule and sachet formulations.

According to the European Summary of Product Characteristics (SmPC), stiripentol dosage escalation should be gradual, starting at 20 mg/kg/day and increasing stepwise depending on age. Dravet syndrome typically begins in infancy, and early initiation of antiepileptic treatment is recommended. A new oral suspension formulation (50 mg/mL) has been developed to facilitate flexible dose adjustments and accurate administration in pediatric patients, especially infants, where precise titration is essential.

This clinical study aims to compare the relative bioavailability of the new oral suspension (test formulation) to the capsule (reference formulation) after a single 1,000 mg dose under fed conditions. In addition to pharmacokinetic endpoints, safety, tolerability, and palatability will be assessed in healthy volunteers. The results will provide critical information on whether the new suspension offers a pharmacokinetic profile comparable to the capsule while improving dosing flexibility and patient convenience in clinical practice.

ELIGIBILITY:
Inclusion Criteria

* Aged between 18 and 50 years (inclusive).
* Considered healthy after a comprehensive clinical assessment (medical history + complete physical exam).
* Body Mass Index (BMI) between 18 and 30 kg/m² (inclusive) and body weight ≥ 50 kg at screening.
* Normal blood pressure (BP) and heart rate (HR) after 10 minutes supine at screening : Systolic BP: 90-145 mmHg, Diastolic BP: 45-90 mmHg, HR: 40-90 bpm, Or values outside these ranges but judged not clinically significant (NCS) by the Investigator.
* Normal ECG at screening (10-min resting 12-lead ECG): PR interval: 110-210 ms, QRS interval : < 120 ms, QTcF interval: ≤ 450 ms, No evidence of sinus node dysfunction, Or values outside these ranges but judged NCS by the Investigator.
* Laboratory parameters within normal ranges (hematology, biochemistry, urinalysis); slight deviations allowed if not clinically relevant per Investigator.
* Women of non-childbearing potential, or women of childbearing potential using at least one acceptable contraceptive method throughout the study and 1 month after last treatment.
* Female subjects of childbearing potential: negative pregnancy test (serum or urine) at screening and Day 0.
* Covered by Health Insurance System and/or compliant with National Law requirements for biomedical research.
* Able and willing to comply with study requirements.
* Written informed consent obtained.

Exclusion Criteria

* Unsuitable veins for repeated venipuncture.
* Relevant history/presence of cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, psychiatric, systemic, or infectious disease.
* Evidence of any clinically significant acute or chronic disease.
* History of suicidal ideation or suicide attempt.
* Surgery (including clinical trial procedures) within 2 months before dosing.
* Blood donation within 2 months before dosing.
* History/presence of drug hypersensitivity, asthma, or allergy.
* Known hypersensitivity to study materials or related compounds.
* Inability/difficulty swallowing capsules.
* No possibility of emergency contact.
* Any drug intake (except paracetamol) within 4 weeks prior to dosing or < 5 half-lives (whichever longer). Prohibited: carbamazepine, phenytoin, phenobarbital, CYP enzyme modulators.
* Use of herbal products affecting CYP enzymes within 2 weeks or < 5 half-lives before dosing.
* Special diets (vegetarian, vegan, gluten-free).
* Vigorous exercise from 4 days before dosing until post-study assessments.
* Pregnant or breastfeeding women.
* Drug/alcohol abuse history, daily alcohol intake > 4 drinks, or positive alcohol test.
* Excessive xanthine beverages (> 5 cups/day).
* Nicotine use > 5 cigarettes/day or inability to abstain 48h before and during study.
* Intake of grapefruit/Seville oranges/poppy seed or other CYP modulators 1 week before dosing and during study.
* Intake of methylxanthines (coffee, tea, cola, cocoa, mate, guarana, chocolate) or quinine (e.g., tonic water) from 48h before dosing and during study.
* Unable/unwilling to follow diet requirements (see protocol section 10.7).
* Positive test for HBsAg, HCV antibody, or HIV 1/2.
* Positive drug screen.
* Significant biological or clinical abnormalities judged incompatible with study.
* Participation in another interventional trial during exclusion period or investigational product within last 60 days or < 5 half-lives.
* Under guardianship, curatorship, or deprived of liberty.
* Under Court protection.
* Would exceed €6000 compensation for biomedical research in last 12 months (including this study).
* Health status not allowing provision of informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability of stiripentol oral suspension (50 mg/mL) vs capsule (500 mg) after a single 1,000 mg oral dose with food, assessed by PK parameters Cmax, AUC0-t, and AUC0-∞ using plasma LC-MS. | Up to 36 hours post-dose (per period)
  The relative bioavailability of stiripentol oral suspension (50 mg/mL) versus capsule (500 mg) after a single 1,000 mg oral dose under fed conditions. It will be assessed by calculating geometric mean ratios with 90% confidence intervals for the main pharmacokinetic parameters: maximum observed plasma concentration (Cmax), area under the concentration-time curve from time zero to the last measurable concentration (AUC0-t), and area under the concentration-time curve extrapolated to infinity (AUC0-∞). Plasma concentrations of stiripentol will be measured using validated liquid chromatography-mass spectrometry (LC-MS) methods to ensure accuracy and reliability of the pharmacokinetic evaluation.

SECONDARY OUTCOMES:
Other PK parameters of stiripentol | Up to 36 hours post-dose (per period).
  Time to maximum concentration (tmax)
Safety and tolerability of stiripentol | From dosing to end of study (~7 weeks per participant).
  Number, nature, incidence, seriousness, severity, and resolution of adverse events following single-dose administration.
Palatability of stiripentol oral suspension | 20 minutes after administration of the oral suspension
  Assessed using a self-administered palatability questionnaire completed 20 minutes after administration of the oral suspension
Other PK parameters of stiripentol | Up to 36 hours post-dose (per period)
  Time before start of absorption (tlag)
Other PK parameters of stiripentol | Up to 36 hours post-dose (per period)
  Elimination rate constant (ke)
Other PK parameters of stiripentol | Up to 36 hours post-dose (per period)
  Terminal half-life (t1/2)
PK parameters of stiripentol metabolites (MIa, MIb) | Up to 36 hours post-dose (per period)
  Maximum concentration (Cmax)
PK parameters of stiripentol metabolites (MIa, MIb) | Up to 36 hours post-dose (per period)
  Area under the curve from time 0 (pre-dose) to the last measurable concentration (AUC0-t)
PK parameters of stiripentol metabolites (MIa, MIb) | Up to 36 hours post-dose (per period)
  Area under the curve from time 0 (pre-dose) to infinity (AUC0-∞)
PK parameters of stiripentol metabolites (MIa, MIb) | Up to 36 hours post-dose (per period)
  Time of occurrence of maximum concentration (tmax)
PK parameters of stiripentol metabolites (MIa, MIb) | Up to 36 hours post-dose (per period)
  Elimination rate constant (ke)
PK parameters of stiripentol metabolites (MIa, MIb) | Up to 36 hours post-dose (per period)
  Apparent terminal elimination half-life (t1/2) measured from plasma concentrations using Liquid chromatography-mass spectrometry (LC-MS)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - 3 Chemin d'Armancourt, Compiègne
  - EUROFINS OPTIMED, 1 rue des Essarts, Gières